CLINICAL TRIAL: NCT06276946
Title: Randomized Assessment of Sparing Parotid Ducts Via MRI Sialography for Reduced Patient-Reported Xerostomia Following Radiotherapy for Oropharynx Cancer
Brief Title: Sparing Parotid Ducts Via MRI Sialography for Reduced Patient Reported Xerostomia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Operational reason
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LCCC2244
Record Dates: First submitted 2024-02-16; First posted 2024-02-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Oropharynx Cancer; Head and Neck Cancer; Xerostomia
Keywords: radiotherapy; magnetic resonance imaging; parotis; parotid duct; radiotherapy dosimetry; radiotherapy planning
MeSH Terms: conditions — Oropharyngeal Neoplasms; Head and Neck Neoplasms; Xerostomia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Mean Parotid (Active Comparator): Standard radiotherapy planning aims to restrict the mean parotid radiation dose to less than or equal to 14 Gy.
  Interventions: Radiation: standard radiotherapy
- Parotid Duct (Experimental): Magnetic resonance images will be used to localize the parotid ducts and limit the radiation dose to these structures to less than or equal to 14 Gy.
  Interventions: Radiation: experimental radiotherapy

INTERVENTIONS:
Radiation: standard radiotherapy — radiotherapy planning goal is to restrict the mean parotid dose is equal to or less than 14Gy.
  Arms: Mean Parotid
Radiation: experimental radiotherapy — radiotherapy planning goal is to restrict the parotid duct dose is equal to or less than 14Gy
  Arms: Parotid Duct

SUMMARY:
Radiation-induced xerostomia (dry mouth) is one of the most common and severe toxicities experienced by patients undergoing radiation treatment for head and neck cancer. Radiation-induced dry mouth is a frequently experienced symptom and persists after treatment, potentially indefinitely. Current practice does not specifically attempt to spare the parotid ducts, where stem/progenitor cells are believed to preferentially reside, and considers the entire salivary gland to have equal function. New radiation therapy planning and conducting strategies are needed to reduce this toxicity and maximize patient quality of life post-treatment.

This randomized Phase II study explores the contribution of magnetic resonance imaging (MRI) guided salivary gland duct definition to decrease patient-reported xerostomia in patients with oropharynx cancer receiving radiation therapy. The severity of xerostomia will be measured by patient-reported (PRO) symptoms, saliva secretion, saliva pH, and buffering.

ELIGIBILITY:
In order to participate in this study a subject must meet all of the eligibility criteria outlined below. Eligibility must be maintained up for the subject to be considered eligible for treatment.

Inclusion Criteria

1. Written informed consent was obtained to participate in the study and HIPAA authorization for the release of personal health information.
2. Subjects is willing and able to comply with study procedures based on the judgment of the investigator.
3. Age ≥ 18 years at the time of consent.
4. T0-4, N0-3, M0 disease American Joint Committee on Cancer (AJCC 7th or 8th edition) of the oropharynx (this includes patients with head and neck cancer of unknown primary origin, often categorized as T0 disease, who will be treated with radiotherapy to the oropharynx) planned for definitive radiotherapy +/- chemotherapy

5 No contraindications to receiving MRI such as implanted electrical devices, pregnancy, and significant quantities of metal in the head/neck

Exclusion Criteria

1. Patients with Sjogren's syndrome or baseline xerostomia (CTCAE > 0 for the question regarding dry mouth)
2. Patients with lesions grossly involving the salivary glands
3. Patients with an allergy to lemon juice
4. Prior history of radiation therapy to the head and neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08-08 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
The difference in patient-reported xerostomia 6 months | 6 months after completion of radiotherapy
  The difference in patient-reported xerostomia will be assessed using the MD Anderson Symptom Inventory -Head & Neck (MDASI-HN) questionnaire. MDASI multi-symptom patient-reported outcome (PRO) measure for clinical and research use. Use the MDASI to assess the severity of symptoms Each question is scaled from 0 to 10. 0= not present and 10= as bad as you imagine.

SECONDARY OUTCOMES:
Saliva mass | 6 months and 12 months after completion of radiotherapy
  The mass of generated saliva post-radiation treatment will be measured.
Parotid duct dose constraint | 6 months after completion of radiotherapy
  The efficacy of 14Gy parotid duct constraint for subjects undergoing parotid ductal sparing radiation therapy will be measured using patient-reported xerostomia scores.
The difference in patient-reported xerostomia 12 months | 12 months after completion of radiotherapy
  The difference in patient-reported xerostomia will be assessed using the MD Anderson Symptom Inventory -Head & Neck (MDASI-HN) questionnaire. MDASI multi-symptom patient-reported outcome (PRO) measure for clinical and research use. Each question is scaled from 0 to 10. 0= not present and 10= as bad as you imagine.
Xerostomia by NCI-CTCAE | 12 months after completion of radiotherapy
  xerostomia will be assessed using The National Cancer Institute Common Terminology Criteria for Adverse Events is a descriptive terminology (NCI-CTCAE) v5.0 that can be utilized for Adverse Event (AE) reporting.
  A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.

CONTACTS AND LOCATIONS:
Overall Officials: Colette Shen, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials